CLINICAL TRIAL: NCT07288970
Title: Comparison of Adductor Canal Block Combined With Sacral Erector Spinae Plane Block Versus Adductor Canal Block Combined With iPACK Block in Patients Undergoing Total Knee Arthroplasty: A Randomized Controlled Tria
Brief Title: ACB With S-ESPB Versus ACB With iPACK for Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study blocks will be performed by an anesthesiologist who is not involved in intraoperative management or postoperative outcome assessment. Study medications and syringes will be prepared by a clinician not involved in patient care. All participants will receive identical appearing syringes, and all blocks will be performed under ultrasound guidance in a standardized fashion. Patients, surgeons, ward staff, investigators, and outcome assessors will remain blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor Canal Block Plus Sacral Erector Spinae Plane Block (ACB + S-ESPB) (Active Comparator): Participants will receive an ultrasound-guided adductor canal block with 20 mL of 0.2% ropivacaine and a sacral erector spinae plane block with 20 mL of 0.2% ropivacaine. All patients will receive standard perioperative care and multimodal analgesia.
  Interventions: Procedure: Adductor Canal Block; Procedure: Sacral Erector Spinae Plane Block
- Adductor Canal Block Plus iPACK Block (ACB + iPACK) (Active Comparator): Participants will receive an ultrasound-guided adductor canal block with 20 mL of 0.2% ropivacaine and an iPACK block with 20 mL of 0.2% ropivacaine. All patients will receive standard perioperative care and multimodal analgesia.
  Interventions: Procedure: Adductor Canal Block; Procedure: iPACK Block

INTERVENTIONS:
Procedure: Adductor Canal Block — Ultrasound-guided adductor canal block performed with 20 mL of 0.2% ropivacaine injected around the saphenous nerve within the adductor canal. Used in both study arms as part of the regional anesthesia protocol for total knee arthroplasty.
  Other Names: ACB
Procedure: Sacral Erector Spinae Plane Block — Ultrasound-guided sacral erector spinae plane block performed with 20 mL of 0.2% ropivacaine injected deep to the erector spinae muscle at the sacral level. Used in combination with ACB in the ACB + S-ESPB group.
  Other Names: S-ESPB; Sacral ESP block
  Arms: Adductor Canal Block Plus Sacral Erector Spinae Plane Block (ACB + S-ESPB)
Procedure: iPACK Block — Ultrasound-guided iPACK block performed with 20 mL of 0.2% ropivacaine injected between the popliteal artery and the posterior capsule of the knee. Used in combination with ACB in the ACB + iPACK group.
  Other Names: Infiltration between the popliteal artery and the posterior capsule of the knee
  Arms: Adductor Canal Block Plus iPACK Block (ACB + iPACK)

SUMMARY:
This study will compare two regional anesthesia strategies for pain management after total knee arthroplasty in adults. Both strategies use an adductor canal block (ACB) to provide analgesia while preserving quadriceps muscle strength. The ACB is then combined with either a sacral erector spinae plane block (S-ESPB) or an iPACK (infiltration between the popliteal artery and the posterior capsule of the knee) block to improve posterior knee analgesia.

All patients will receive an ultrasound-guided adductor canal block with 20 mL of 0.2% ropivacaine. They will then be randomly assigned to one of two groups:

Group 1: ACB combined with a sacral erector spinae plane block (S-ESPB) using 20 mL of 0.2% ropivacaine.

Group 2: ACB combined with an iPACK block using 20 mL of 0.2% ropivacaine. Both techniques aim to provide effective postoperative analgesia while minimizing motor blockade and allowing for early mobilization. It is not known whether combining ACB with S-ESPB or with iPACK provides superior pain control, reduces opioid requirements, or results in better functional recovery after total knee arthroplasty.

The main purpose of this study is to compare the time to first rescue analgesia and overall postoperative pain control between the two regional anesthesia strategies. The study will also evaluate opioid consumption, motor function, functional mobility, side effects, and block-related complications.

We hypothesize that both combinations will provide effective analgesia, but their impact on pain intensity, duration of analgesia, and functional recovery may differ.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is associated with significant postoperative pain, which can limit early mobilization, delay rehabilitation, and increase opioid use. Inadequate pain control may lead to complications such as decreased range of motion, prolonged hospitalization, and reduced patient satisfaction. Regional anesthesia techniques are a cornerstone of multimodal analgesia protocols for TKA.

The adductor canal block (ACB) is a motor-sparing technique that targets the saphenous nerve and nerve to vastus medialis while largely preserving quadriceps strength. However, ACB alone may not provide sufficient analgesia for posterior knee structures. To address this limitation, it is often combined with other blocks that target posterior knee innervation.

The iPACK (infiltration between the popliteal artery and the posterior capsule of the knee) block is designed to anesthetize the articular branches supplying the posterior capsule of the knee without causing significant motor block. The sacral erector spinae plane block (S-ESPB) is a more proximal truncal block, which may provide analgesia to the posterior knee and surrounding structures through spread of local anesthetic in the fascial planes.

This randomized controlled trial will compare two regional anesthesia strategies in patients undergoing total knee arthroplasty:

Adductor canal block (ACB) combined with sacral erector spinae plane block (S-ESPB).

Adductor canal block (ACB) combined with iPACK block. In both groups, 20 mL of 0.2% ropivacaine will be used for each block (ACB + S-ESPB or ACB + iPACK). All patients will receive standard perioperative care and multimodal analgesia according to institutional protocols.

The primary outcome of the study is the time to first rescue analgesia within 48 hours after surgery. Secondary outcomes include pain intensity at rest and during movement, total opioid consumption, motor function (quadriceps strength), postoperative nausea and vomiting, hemodynamic events, block-related complications, time to first mobilization, and patient satisfaction with pain management.

The study aims to determine whether combining ACB with S-ESPB or with iPACK results in better analgesia and functional outcomes after TKA. The results may help optimize regional anesthesia protocols for total knee arthroplasty and improve postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Scheduled for elective unilateral total knee arthroplasty under spinal or general anesthesia
* ASA physical status I-III
* Planned use of regional anesthesia with an adductor canal block as part of multimodal analgesia
* Ability to communicate pain intensity using the NRS scale
* Written informed consent obtained from the patient

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Allergy, intolerance, or contraindication to local anesthetics (ropivacaine)
* Pre-existing significant neurological deficit or neuropathy in the operative limb
* Coagulopathy or anticoagulation that contraindicates peripheral nerve blocks (e.g., INR >1.5, platelets <100,000/µL, or therapeutic anticoagulation that cannot be safely paused)
* Infection at or near the planned needle insertion sites
* Severe hepatic or renal impairment
* Chronic opioid therapy (>30 days of daily opioid use before surgery)
* Cognitive impairment or delirium preventing reliable pain assessment BMI > 40 kg/m² (optional - if chcesz ograniczyć ze względu na trudność USG)
* Previous knee arthroplasty on the same side or revision TKA (jeśli chcesz tylko primary TKA)
* Pregnancy or breastfeeding
* Participation in another interventional clinical trial within 30 days

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to First Rescue Analgesia | Within 48 hours after surgery.
  Time (in hours) from completion of the regional blocks to the first administration of a rescue analgesic (opioid or non-opioid) given for pain intensity ≥4 on the 0-10 Numerical Rating Scale (NRS).

SECONDARY OUTCOMES:
Pain Intensity at Rest (NRS 0-10) | 4 hours after surgery.
  Pain at rest measured using the 0-10 NRS (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 8 hours after surgery.
  Pain at rest measured using the 0-10 NRS (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 12 hours after surgery.
  Pain at rest measured using the 0-10 NRS (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 24 hours after surgery.
  Pain at rest measured using the 0-10 NRS (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 48 hours after surgery.
  Pain at rest measured using the 0-10 NRS (0 = no pain, 10 = worst imaginable pain). Mean values will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 4 hours after surgery.
  Pain during standardized knee movement (e.g., flexion or assisted mobilization) measured using the 0-10 NRS.
Pain Intensity During Movement (NRS 0-10) | 8 hours after surgery.
  Pain during standardized knee movement (e.g., flexion or assisted mobilization) measured using the 0-10 NRS.
Pain Intensity During Movement (NRS 0-10) | 12 hours after surgery.
  Pain during standardized knee movement (e.g., flexion or assisted mobilization) measured using the 0-10 NRS.
Pain Intensity During Movement (NRS 0-10) | 24 hours after surgery.
  Pain during standardized knee movement (e.g., flexion or assisted mobilization) measured using the 0-10 NRS.
Pain Intensity During Movement (NRS 0-10) | 48 hours after surgery.
  Pain during standardized knee movement (e.g., flexion or assisted mobilization) measured using the 0-10 NRS.
Total Opioid Consumption | 0-48 hours after surgery.
  Cumulative dose of opioids converted to oral morphine milligram equivalents (MME).
Motor Function (Quadriceps Strength, MRC Scale) | 4 hours after surgery.
  Quadriceps muscle strength assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the regional anesthesia techniques.
Motor Function (Quadriceps Strength, MRC Scale) | 8 hours after surgery.
  Quadriceps muscle strength assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the regional anesthesia techniques.
Motor Function (Quadriceps Strength, MRC Scale) | 12 hours after surgery.
  Quadriceps muscle strength assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the regional anesthesia techniques.
Motor Function (Quadriceps Strength, MRC Scale) | 24 hours after surgery.
  Quadriceps muscle strength assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the regional anesthesia techniques.
Motor Function (Quadriceps Strength, MRC Scale) | 48 hours after surgery.
  Quadriceps muscle strength assessed using the Medical Research Council (MRC) scale (0 = no contraction; 5 = normal power) to detect any motor impairment associated with the regional anesthesia techniques.
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-48 hours after surgery.
  Presence of nausea or vomiting requiring antiemetic therapy. Proportion of patients with at least one episode will be recorded.
Hemodynamic Adverse Events | From block placement until 24 hours after surgery.
  Incidence of hypotension (systolic BP <90 mmHg or >30% decrease from baseline) and bradycardia (HR <50/min) requiring treatment.
Block-Related Adverse Events | From block placement until 30 days after surgery.
  Incidence of complications related to the regional blocks, including prolonged sensory or motor deficit, nerve injury (evaluated in outpatient clinic if required), hematoma, infection at the injection site, persistent weakness, or local anesthetic systemic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, MD PhD, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after publication, available for 5 years
Access Criteria: upon reasonable request; de-identified data; DSA if needed